CLINICAL TRIAL: NCT03828539
Title: Head-to-head Study of Erenumab Against topiRamate-a Double-blind, Double Dummy Migraine Study to Assess Tolerability and Efficacy in a patiEnt -Centered Setting
Brief Title: Head-to-head Study of Erenumab Against Topiramate in Patients With Episodic and Chronic Migraine
Acronym: HER-MES
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CAMG334ADE01; 2018-000943-15 (EudraCT Number)
Record Dates: First submitted 2019-02-01; First posted 2019-02-04 (Actual); Results first posted 2021-08-09 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Migraine
Keywords: Migraine; Episodic migraine; Chronic migraine; Headache; erenumab; topiramate; CAMG 334; Calcitonin Gene-related Peptide; CGRP; CGRP receptor agonist; monoclonal antibody; treatment failure
MeSH Terms: conditions — Migraine Disorders; Headache | interventions — erenumab; Topiramate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Erenumab (Experimental): 70 mg and 140 mg Erenumab
  Interventions: Biological: Erenumab; Biological: Erenumab matching placebo
- Topiramate (Active Comparator): Topiramate in the highest tolerated dose (50 - 100 mg/day)
  Interventions: Drug: Topiramate; Drug: Topiramate matching placebo

INTERVENTIONS:
Biological: Erenumab — 70mg/1mL (70 mg) or 2x70mg/1mL (140 mg) in pre-filled syringe, administered every 4 weeks
  Other Names: AMG334
  Arms: Erenumab
Drug: Topiramate — Film-coated tablet taken orally:
  25 mg administered once daily (first week of titration phase). After the first week, titration was done according to the summary of product characteristics (SmPC) in 25 mg increments each week and aimed to reach the recommended daily treatment dose of 100 mg (50/75/100 mg). 50/75/100 mg were administered twice daily during titration phase and maintenance phase.
  Other Names: Topamax
  Arms: Topiramate
Biological: Erenumab matching placebo — Erenumab matching placebo pre-filled syringue administered every 4 weeks
  Arms: Erenumab
Drug: Topiramate matching placebo — Topiramate matching placebo administered daily
  Arms: Topiramate

SUMMARY:
This study used a single-cohort, 2-treatment arm, parallel-group randomized, double-blind, double-dummy design in adult patients with episodic migraine and chronic migraine, who had to be either naïve or not suitable for or could have failed up to three prophylactic treatments out of: propranolol/metoprolol, amitriptyline, flunarizine. Patients were stratified into groups according to their number of migraine days during the baseline period.

DETAILED DESCRIPTION:
All patients completing the Baseline period and fulfilling baseline eligibility criteria were invited to participate to the Double-blind, double-dummy Treatment Epoch (DBTE, 24 weeks) .

Eligible patients were randomized to one of two treatment arms. DBTE started with a titration phase for topiramate of a maximum of 6 weeks to determine the maximal tolerated dose and aimed to reach the recommended treatment dose of 100 mg according to the German SmPC. After the titration phase, maintenance phase started (18 weeks). Topiramate dose had to be maintained until the end of the DBTE. Erenumab dose at beginning of the DBTE was determined patient individually by the investigator based on the guidance provided in the SmPC and was either 70 mg or 140 mg. Dose escalation from 70 mg to 140 mg in case of insufficient response was considered at anytime during the DBTE.

Dose reduction of topiramate and erenumab was not allowed during DBTE (Week 0 to Week 24). After Week 24 or if the patient discontinued study drug, a one week double-blind taper off phase followed to ensure proper down titration for topiramate. At the end of the DBTE (24 weeks) the final assessment occurred to address the objectives.

A Follow-Up Visit 4 weeks after last study visit (or 8 weeks after last IMP injection for discontinued patients) was required as part of routine safety monitoring. The primary analysis was triggered when all patients had completed their respective last visit of the DBTE.

The End of study occurred when the last patient completed last visit (LPLV).

ELIGIBILITY:
Key Inclusion Criteria:

1. Documented history of migraine in the 12 months prior to screen
2. at least 4 days per month of migraine symptoms
3. >=80% diary compliance during the Baseline period
4. Patients must be either naïve or not suitable or have failed previous migraine prophylactic treatments

Key Exclusion Criteria:

1. Older than 50 years of age at migraine onset
2. Pregnant or nursing
3. History of cluster or hemiplegic headache
4. History or evidence of major psychiatric disorder
5. Score of 19 or higher on Beck Depression Inventory (BDI)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 777 (Actual)
Dates: Start 2019-02-22 (Actual); Primary Completion 2020-07-29 (Actual); Study Completion 2020-07-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (64):
- Germany (64):
  - Novartis Investigative Site, Stuttgart, Baden-Wurttemberg
  - Novartis Investigative Site, Marburg Wehrda, Germany
  - Novartis Investigative Site, Hanover, Lower Saxony
  - Novartis Investigative Site, Aachen, North Rhine-Westphalia
  - Novartis Investigative Site, Alzenau in Unterfranken
  - Novartis Investigative Site, Bad Homburg
  - Novartis Investigative Site, Bad Honnef
  - Novartis Investigative Site, Bad Saarow
  - Novartis Investigative Site, Bayreuth
  - Novartis Investigative Site, Bergen
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bielefeld
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Böblingen
  - Novartis Investigative Site, Celle
  - Novartis Investigative Site, Chemnitz
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Dillingen
  - Novartis Investigative Site, Erbach im Odenwald
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Gelsenkirchen
  - Novartis Investigative Site, Greifswald
  - Novartis Investigative Site, Haar
  - Novartis Investigative Site, Halle
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Heidenheim
  - Novartis Investigative Site, Hoppegarten
  - Novartis Investigative Site, Ibbenbueren
  - Novartis Investigative Site, Jena
  - Novartis Investigative Site, Jülich
  - Novartis Investigative Site, Kassel
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Königstein im Taunus
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Lünen
  - Novartis Investigative Site, Mannheim
  - Novartis Investigative Site, Mittweida
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Neu-Ulm
  - Novartis Investigative Site, Neuburg an der Donau
  - Novartis Investigative Site, Osnabrück
  - Novartis Investigative Site, Pforzheim
  - Novartis Investigative Site, Quakenbrück
  - Novartis Investigative Site, Regensburg
  - Novartis Investigative Site, Rostock
  - Novartis Investigative Site, Rülzheim
  - Novartis Investigative Site, Schwerin
  - Novartis Investigative Site, Seesen
  - Novartis Investigative Site, Siegen
  - Novartis Investigative Site, Sindelfingen
  - Novartis Investigative Site, Stadtroda
  - Novartis Investigative Site, Stuttgart
  - Novartis Investigative Site, Trier
  - Novartis Investigative Site, Tübingen
  - Novartis Investigative Site, Ulm
  - Novartis Investigative Site, Unterhaching
  - Novartis Investigative Site, Westerstede/Oldenburg
  - Novartis Investigative Site, Wiesbaden
  - Novartis Investigative Site, Würzburg

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Ehrlich M, Hentschke C, Sieder C, Maier-Peuschel M, Reuter U. Erenumab versus topiramate: post hoc efficacy analysis from the HER-MES study. J Headache Pain. 2022 Nov 15;23(1):141. doi: 10.1186/s10194-022-01511-y. PMID 36380284
- [Derived] Reuter U, Ehrlich M, Gendolla A, Heinze A, Klatt J, Wen S, Hours-Zesiger P, Nickisch J, Sieder C, Hentschke C, Maier-Peuschel M. Erenumab versus topiramate for the prevention of migraine - a randomised, double-blind, active-controlled phase 4 trial. Cephalalgia. 2022 Feb;42(2):108-118. doi: 10.1177/03331024211053571. Epub 2021 Nov 7. PMID 34743579
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=941

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 82 centers in Germany enrolled patients.
Pre-assignment Details: A total of 777 patients were randomized to receive either erenumab (389 patients) or topiramate (388 patients).
Period: Overall Study
Arm/Group | Erenumab | Topiramate
Started (All patients who received a randomization number, regardless of receiving study medication were included in the Randomized Set) | 389 | 388
Full Analysis Set (FAS) (All patients who received at least one dose of active study medication. In FAS, patients were analyzed according to randomized treatment, regardless of the actual treatment received.) | 388 | 388
Safety Analysis Set (SAF) (All randomized patients who received at least one dose of active study medication. In the SAF, patients were analyzed based on actual treatment received.) | 388 | 388
Completed | 373 | 366
Not Completed | 16 | 22
Not completed — Adverse Event | 3 | 12
Not completed — Patient's/guardian's decision | 3 | 5
Not completed — Lost to Follow-up | 4 | 2
Not completed — Protocol Violation | 3 | 2
Not completed — Withdrawal of informed consent | 2 | 1
Not completed — New therapy for study indication | 1 | 0

BASELINE CHARACTERISTICS:
Population: Demographic variables and other baseline characteristics were summarized for each randomized treatment group and for all patients (total) using the Full Analysis set (FAS)
Groups:
- Total: Total of all reporting groups
Arm/Group | Erenumab | Topiramate | Total
Number analyzed (Participants) | 388 | 388 | 776
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.8 (12.4) | 40.7 (12.4) | 40.7 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 331 | 335 | 666
  Male | 57 | 53 | 110
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 383 | 387 | 770
  Asian | 1 | 0 | 1
  Unknown | 1 | 0 | 1
  Other | 3 | 1 | 4
Baseline Monthly Migraine Days (MMDs) categories [Count of Participants; unit: Participants] — Monthly migraine days at baseline are the number of migraine days in the baseline period that are normalized in a 28-day interval. Monthly migraine days after baseline are the number of migraine days between each monthly IMP dose that are normalized in a 28-day interval. Days without eDiary data in each normalized monthly interval were prorated.
  Participants
    < 4 days | 2 | 0 | 2
    4 to 7 days | 94 | 92 | 186
    8 to 14 days | 248 | 254 | 502
    >= 15 days | 43 | 42 | 85
    Missing | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Treatment Discontinuation Due to an Adverse Event (AE) During the Double-blind Treatment Epoch/Period (DBTE)
Description: The primary objective was to demonstrate the tolerability of 70 mg and 140 mg erenumab compared to topiramate in the highest tolerated dose assessed by the rate of patients discontinuing treatment due to AE during the double-blind epoch of the study.
Time Frame: 24 Weeks
Population: Full Analysis Set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | Erenumab | Topiramate
Number analyzed (Participants) | 388 | 388
Participants | 41 | 151
Statistical Analysis 1: Comparison: Erenumab vs Topiramate; Test type: Other; p < .001, Regression, Logistic; Odds ratio is obtained from a logistic regression model that includes treatment group and stratification factor (MMD at baseline); Odds Ratio (OR) = 0.19, 95% CI 2-sided [0.13 to 0.27]

2. Secondary Outcome: Number of Patients With at Least 50% Reduction From Baseline in Monthly Migraine Days (MMD) Over the Last Three Months (Month 4, 5, and 6)
Description: The secondary objective of this study was to evaluate the effect of erenumab compared to topiramate on the proportion of patients with at least 50% reduction from baseline in MMDs. The Baseline period was defined as the period between Week -4 and the day prior to first dose. This was analyzed by logistic regression over the last 3 months (months 4, 5, and 6) of treatment. All the subjects' data collected regarding 50% response in MMD was used in the analysis regardless of whether subjects discontinue study treatment or not. Subjects with missing response information on this endpoint were imputed as non-response (non-responder imputation).
Time Frame: Baseline, Last three months (month 4, 5, and 6)
Population: Full Analysis Set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | Erenumab | Topiramate
Number analyzed (Participants) | 388 | 388
Participants | 215 | 121
Statistical Analysis 1: Comparison: Erenumab vs Topiramate; Test type: Other; p < .001, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 2.76, 95% CI 2-sided [2.06 to 3.71]

3. Other Pre Specified Outcome: EXPLORATORY ENDPOINT: Proportion of Patients Achieving at Least a 5 Points Reduction in the Headache Impact Test (HIT-6) From Baseline to Week 24
Description: The HIT-6 is a widely used patient-reported outcome measure that assesses the negative effects of headaches on normal activity. Six items assess the frequency of pain severity, headaches limiting daily activity (household, work, school, and social), wanting to lie down when headache is experienced, feeling too tired to work or do daily activities because of headache, feeling "fed up" or irritated because of headache, and headaches limiting ability to concentrate or work on daily activities. Each of the 6 questions is responded to using 1 of 5 response categories: "never," "rarely," "sometimes," "very often," or "always." For each HIT-6 item, 6, 8, 10, 11, or 13 points, respectively, are assigned to the response provided. These points are summed to produce a total HIT-6 score that ranges from 36 to 78. HIT-6 scores are categorized into 4 grades: little or no impact (49 or less), some impact (50 - 55), substantial impact (56 - 59), and severe impact (60 - 78) due to headache.
Time Frame: Baseline, Week 24
Population: Full Analysis Set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | Erenumab | Topiramate
Number analyzed (Participants) | 388 | 388
Participants | 280 | 209
Statistical Analysis 1: Comparison: Erenumab vs Topiramate; Test type: Other; p < .001, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 2.30, 95% CI 2-sided [1.70 to 3.12]

4. Other Pre Specified Outcome: EXPLORATORY ENDPOINT: Proportion of Patients Achieving at Least a 5 Points Increase in the Medical Outcome Short Form Health Survey Version 2 (SF-36) From Baseline to Week 24
Description: The SF-36 is a widely used and extensively studied instrument to measure health-related quality of life (HRQoL) among healthy subjects and patients with acute and chronic conditions. It consists of eight subscales that can be scored individually: Physical Functioning, Role-Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role-Emotional, and Mental Health. Two overall summary scores, the Physical Component Summary (PCS) and the Mental Component Summary (MCS) also can be computed. The SF-36 has proven useful in monitoring general and specific populations, comparing the relative burden of different disease, differentiating the health benefits produced by different treatments, and in screening individual patients. The purpose of the SF-36 in this study was to assess the HRQoL of patients. Given the nature of this disease and the 4-weekly assessment, the SF-36 version 2, with a 4-week recall period, was used in this study.
Time Frame: Baseline, Week 24
Population: Full Analysis Set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | Erenumab | Topiramate
Number analyzed (Participants) | 388 | 388
Participants
  Physical Component Summary (PCS) | 185 | 145
  Mental Component Summary (MCS) | 98 | 65
Statistical Analysis 1: Comparison: Erenumab vs Topiramate; Physical Component Summary (PCS); Test type: Other; p < 0.001, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.75, 95% CI 2-sided [1.26 to 2.43]
Statistical Analysis 2: Comparison: Erenumab vs Topiramate; Mental Component Summary (MCS); Test type: Other; p = 0.005, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.79, 95% CI 2-sided [1.29 to 2.69]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment until 8 weeks after the last Investigational Medicinal product (IMP) injection, assessed up to approximately 33 weeks (treatment duration ranged from 4.0 to 25.1 weeks).
Description: Any sign or symptom that occurs during the study treatment until 8 weeks after the last Investigational Medicinal product (IMP) injection. Maximum exposure to study treatments = 25 weeks (Erenumab treatment group) and 25.1 weeks (Topiramate treatment group).
Arm/Group | Erenumab | Topiramate
All-Cause Mortality (participants affected / at risk) | 0/388 | 0/388
Serious Adverse Events (participants affected / at risk) | 10/388 | 19/388
Other Adverse Events (participants affected / at risk) | 253/388 | 331/388
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erenumab (N=388) | Topiramate (N=388)
Angle closure glaucoma (Eye disorders) | 0 | 1
Retinal detachment (Eye disorders) | 0 | 1
Rhegmatogenous retinal detachment (Eye disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 1
Mechanical ileus (Gastrointestinal disorders) | 1 | 0
Obstructive defaecation (Gastrointestinal disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Anaphylactic shock (Immune system disorders) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1
Bacteriuria (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Gastrointestinal infection (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1
Papilloma viral infection (Infections and infestations) | 1 | 0
Parasitic gastroenteritis (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0
Sternal fracture (Injury, poisoning and procedural complications) | 1 | 0
Tendon injury (Injury, poisoning and procedural complications) | 1 | 0
Weight decreased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Migraine (Nervous system disorders) | 0 | 1
Migraine with aura (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Major depression (Psychiatric disorders) | 1 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0
Endometriosis (Reproductive system and breast disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Erenumab (N=388) | Topiramate (N=388)
Vertigo (Ear and labyrinth disorders) | 20 | 24
Abdominal pain upper (Gastrointestinal disorders) | 22 | 23
Constipation (Gastrointestinal disorders) | 48 | 12
Diarrhoea (Gastrointestinal disorders) | 20 | 29
Nausea (Gastrointestinal disorders) | 36 | 71
Fatigue (General disorders) | 44 | 74
Nasopharyngitis (Infections and infestations) | 145 | 150
Weight decreased (Investigations) | 5 | 22
Decreased appetite (Metabolism and nutrition disorders) | 8 | 39
Back pain (Musculoskeletal and connective tissue disorders) | 21 | 20
Disturbance in attention (Nervous system disorders) | 18 | 63
Dizziness (Nervous system disorders) | 28 | 60
Dysgeusia (Nervous system disorders) | 3 | 23
Paraesthesia (Nervous system disorders) | 17 | 159
Taste disorder (Nervous system disorders) | 0 | 26
Sleep disorder (Psychiatric disorders) | 20 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-06-06): https://cdn.clinicaltrials.gov/large-docs/39/NCT03828539/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-01): https://cdn.clinicaltrials.gov/large-docs/39/NCT03828539/SAP_001.pdf